CLINICAL TRIAL: NCT00231556
Title: A Randomized, Double-Blind, Parallel-Group, Monotherapy Study to Compare the Safety and Efficacy of Two Doses of Topiramate in the Treatment of Newly Diagnosed or Recurrent Epilepsy
Brief Title: A Study on Safety and Efficacy of Two Doses of Topiramate as Monotherapy in the Treatment of Newly Diagnosed or Recurrent Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003259
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-01

CONDITIONS: Epilepsy; Seizures; Epilepsies, Partial; Epilepsy, Generalized; Epilepsy, Tonic-Clonic
Keywords: Epilepsy; Seizures; Parital Epilepsies; Generalized Epilepsy; Tonic-Clonic Epilepsy; Topiramate
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial; Epilepsy, Generalized; Epilepsy, Tonic-Clonic | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two doses of topiramate as monotherapy in the treatment of pediatric and adult patients with newly diagnosed or recurrent epilepsy.

DETAILED DESCRIPTION:
Topiramate is approved for treating epilepsy in combination with other epilepsy drugs, but not approved for treating epilepsy as sole treatment or in recently diagnosed epilepsy characterized by partial-onset seizures. This is a randomized, double-blind, parallel-group, multicenter study to compare the safety and effectiveness of two doses of topiramate as monotherapy in pediatric and adult patients with newly diagnosed (within 3 months) or recurrent epilepsy (partial-onset or primary generalized tonic-clonic). The study consists of 4 phases: Baseline (assessment of seizure frequency and other eligibility), Open-Treatment (all patients receive 25 milligrams[mg]/day of topiramate for 7 days), Core Double-Blind Phase (patients are randomized to receive either their assigned dose of topiramate of 50mg/day or 400mg/day, or maximum tolerated dose, and then remain, if possible, on that dose for the duration of the double-blind phase; they continue to receive the medication until they experience the first seizure or until 6 months after the last patient is enrolled), and Long-Term Extension Phase (patients continue to receive the medication at maximum tolerated dose, which may be adjusted according to individual tolerability and effectiveness, until either the patient withdraws or the sponsor terminates the study). The study hypothesis is that topiramate will be effective in the treatment of newly diagnosed or recurrent epilepsy in dose-dependent manner. Topiramate tablets (25 milligrams[mg]) daily by mouth in once-daily regimen during the 7-day Open-Treatment Phase; topiramate twice daily for total of 50mg/day or 400mg/day during the Double-Blind Phase.

ELIGIBILITY:
Inclusion Criteria:

* Weigh >=25 kilograms
* Diagnosis of epilepsy within 3 months prior to study entry or recurrence of epilepsy while off of anit-epileptic drugs
* No more than two documented seizures during the three-month retrospective baseline phase
* may have experienced seizures prior to the three-month, retrospective baseline phase
* Patients with partial-onset seizures, with or without a secondarily generalized component, and generalized seizures, including tonic-clonic (grand mal), tonic, clonic, juvenile myoclonic epilepsy (impulsive petit mal) and myoclonic epilepsy
* Receiving either no other concomitant anti-epileptic drug (AED) or be on one standard AED.

Exclusion Criteria:

* Patients who do not have epilepsy
* Patients with absence (petit mal) or atypical absence seizures, epilepsia paritlis continua, cluster pattern or serial seizures
* Patients with progressive neurological or degenerative disorder
* Patients with significant history of unstable medical diseases
* Patients with a drug allergy or hypersensitivity to carbonic anhydrase inhibitors or sulfa drugs
* Patients with history of alcohol or drug abuse within past one year
* Patients with a history of suicide attempt within past one year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 1999-07; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Time to first seizure (partial onset or generalized tonic-clonic seizure) during the core double-blind phase (excluding taper).

SECONDARY OUTCOMES:
Mean plasma topiramate levels for the high and low topiramate dosing groups; laboratory evaluations, vital signs, visual field testing results, and adverse events during trial

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study on Safety and Efficacy of Two Doses of Topiramate as Monotherapy in the Treatment of Newly Diagnosed or Recurrent Epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=516&filename=CR003259_CSR.pdf